CLINICAL TRIAL: NCT01429194
Title: Continuation of Follow-up for Patients Who Were Previously Enrolled in the Clinical Study: "Open Prospective Study to Evaluate the Safety and Preliminary Effectiveness of the BaroSense ACE Stapler for the Treatment of Obesity - (Protocol 11-03)."
Brief Title: The ACE Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90891629; 90891629 (Other: Boston Scientific Corporation)
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: Weight Loss; Trans-oral Endoscopic Procedure; Gastric Plication
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACE procedure (Experimental): ACE procedure for the treatment of obesity
  Interventions: Procedure: ACE Stapler

INTERVENTIONS:
Procedure: ACE Stapler — The ACE Stapler is used endoscopically, and incorporates a unique tissue capture mechanism to produce large, permanent serosa to serosa plications in a completely trans-oral approach.

SUMMARY:
The Articulating Circular Endoscopic (ACE) Stapler is an investigational system using endoscopic guidance to trans-orally place plications in the stomach in obese subjects to reduce volume and expansion of the fundus and greater curve to abate hunger as part of a supervised weight reduction program.

The primary objective of this study is to perform an evaluation of the safety of the plication procedure.

The secondary objective of this study is to evaluate the preliminary efficacy of the ACE Stapler for the treatment of obesity over a 24 month follow-up period.

DETAILED DESCRIPTION:
This study was originally sponsored by BaroSense, Inc (protocol 11-03). 69 subjects were enrolled and treated as part of the study at 6 centers in 4 countries outside the United States. On April 30, 2013 BaroSense Inc went out of business and the study was terminated with all participating centers' Ethics Committees. At the point of study termination, all patients were in the middle of post procedure follow-up.

Boston Scientific has since acquired the technology and study and will re-initiate follow-up to 24 months in order to collect data to support the original safety and efficacy endpoints of the protocol. Only the 69 subjects previously enrolled and treated in BaroSense's protocol 11-03 will be eligible for participation in the Boston Scientific continued follow-up study ("The ACE Follow-up Study" protocol 90891629). The Boston Scientific protocol will be approved by participating centers' Ethics Committees and patients who choose to participate in The ACE Follow-up Study will need to sign a new, Ethics Committee Approved, informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Subject, male or female, is age 18 to 50 years of age.
2. Subject must be able to understand and be willing to sign an informed consent document.
3. Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study. This includes availability of reliable transportation and sufficient time to attend all follow-up visits.
4. Subject has a BMI of 40 - 45 or 30 to 39.9 plus one or more co-morbid diseases expected to improve with weight loss, including but not limited to hypertension, dyslipidemia, obstructive sleep apnea, or diabetes mellitus.
5. Subject must be fully ambulatory, without chronic reliance on walking aids such as crutches, walkers or a wheelchair.
6. Subject must be of sufficient and stable medical health, as evaluated by the Principal Investigator.
7. Subject must have a primary care physician that will manage the subject for any co-morbid conditions throughout the study.
8. Subject must have failed standard obesity therapy of diet, exercise, behavior modification, and pharmacologic agents either alone or in combination, as assessed by an interview with a member of the study team at baseline.
9. Subject agrees to refrain from any type of reconstructive surgery that may affect body weight such as mammoplasty or abdominal lipoplasty or liposuction, during the trial.

Exclusion Criteria:

1. Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease.
2. Subject has poorly controlled diabetes as indicated by the lack of stable diabetes medications and doses over the last month, or has a history of diabetes for greater than 10 years.
3. Subject has had significant weight loss in the last 3 months, or between baseline and the study procedure.
4. Subject has a history or is diagnosed with eating disorders.
5. Subject has history of peptic ulcer and tests positive for H. pylori, unless treated before the procedure.
6. Subject has symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
7. Subject has pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
8. Subject has significant esophageal disease including Zenker's diverticulum, grade 3-4 reflux esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, or symptoms of dysmotility.
9. Subject is observed during EGD to have heavily scarred, malignant or poor quality/friable tissue in areas of the stomach where plications are to be placed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety | Enrollment through 24 months post-procedure.
  The primary safety analysis will assess the occurrence and procedure relatedness of the following events:
  * Adverse Events (AE)
  * Adverse Device Effects (ADE)
  * Serious Adverse Events (SAE)
  * Unanticipated Adverse Device Effects (UADE)

SECONDARY OUTCOMES:
Percent excess weight loss | Procedure through 24 months post-procedure
  Percent excess weight loss (%EWL), defined as: (preoperative weight-current weight)/(preoperative weight - ideal weight) *100, where ideal weight is the weight that would correspond to a BMI of 25 based on the subject's height.
  Relative to weight at the procedure visit.
Total weight lost (kg) and percent weight lost | Procedure through 24 months post-procedure
  Relative to weight at the procedure visit.
Change in Body Mass Index (BMI) and percent change in BMI | Procedure through 24 months post-procedure
  Relative to BMI at the procedure visit.
Change in waist circumference | Procedure through 24 months post-procedure
  Relative to to waist circumference at the procedure visit.
Improvement in co-morbid disease(s) | Enrollment through 24 months post-procedure
  Including but not limited to, improvement in vital signs and/or laboratory values.
Changes in Quality of Life | Enrollment through 24 months post-procedure
  As reported on the SF-36 Quality of LIfe Questionnaire.
Changes in Feelings of Satiety | Enrollment through 24 months post-procedure
  As reported on the TFEQ-R18 Three Factor Eating Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Biron, MD, Principal Investigator — University Institute of Cardiology and Pulmonary Medicine of Quebec
Locations (6):
- Argentina (2):
  - Hospital Aleman / Programa de Unidades Bariátricas, Autonoma de Bueno Aires
  - Hospital Italiano de Mendoza / Clinica Quirugica S. A., Mendoza
- University Institute of Cardiology and Pulmonary Medicine of Quebec, Québec, Quebec, Canada
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel
- Netherlands (2):
  - Amsterdam Medical Center, Amsterdam
  - University Hospital Maastricht, Maastricht

REFERENCES:
- [Derived] Verlaan T, Paulus GF, Mathus-Vliegen EM, Veldhuyzen EA, Conchillo JM, Bouvy ND, Fockens P. Endoscopic gastric volume reduction with a novel articulating plication device is safe and effective in the treatment of obesity (with video). Gastrointest Endosc. 2015 Feb;81(2):312-20. doi: 10.1016/j.gie.2014.06.017. Epub 2014 Jul 29. PMID 25085333